CLINICAL TRIAL: NCT01207271
Title: A Comparison of Cognitive and Dynamic Therapy for MDD in Community Settings
Brief Title: A Comparison of Cognitive and Dynamic Therapy for Depression in Community Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01HS018440 (AHRQ)
Record Dates: First submitted 2010-09-21; First posted 2010-09-22 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Major Depressive Disorder
Keywords: depression; community mental health; treatment; psychotherapy; mediators
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Cognitive Behavioral Therapy; Psychotherapy, Psychodynamic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Therapy (Experimental)
  Interventions: Behavioral: Cognitive Therapy
- Dynamic Therapy (Experimental)
  Interventions: Behavioral: Supportive-Expressive Psychodynamic Therapy

INTERVENTIONS:
Behavioral: Cognitive Therapy — 16 sessions of cognitive therapy administered weekly by a community mental health therapist
  Other Names: Cognitive Behavioral Therapy; CBT
  Arms: Cognitive Therapy
Behavioral: Supportive-Expressive Psychodynamic Therapy — 16 sessions of supportive-expressive psychodynamic therapy administered weekly by a community mental health therapist
  Other Names: Psychodynamic Psychotherapy; Short Term Dynamic Therapy
  Arms: Dynamic Therapy

SUMMARY:
The goal of this study is to compare supportive-expressive therapy, a type of psychodynamic psychotherapy, with cognitive therapy for the treatment of depression in community mental health consumers.

Hypothesized mediators of treatment will also be examined.

DETAILED DESCRIPTION:
The goal of this study is to conduct a randomized, comparative, non-inferiority clinical trial that tests the hypothesis that a widely used form of manualized dynamic psychotherapy (supportive-expressive psychodynamic therapy) is not inferior to cognitive therapy when implemented in community mental health settings for the treatment of major depressive disorder (MDD). The specific aims are (1) to conduct a randomized non-inferiority trial to compare supportive-expressive psychodynamic therapy and cognitive therapy for patients with MDD and (2) to assess the comparative effectiveness of supportive-expressive psychodynamic therapy and cognitive therapy on secondary measures of symptoms, patient functioning, and quality of life.

Patient mediators of outcome will also be examined through an additional grant awarded to Paul Crits-Christoph, Ph.D. This grant was funded by the National Institutes of Mental Health - RO1MH092363-01. This grant is entitled:"The mechanisms of cognitive and dynamic therapy in community settings."

Recruitment will occur solely through community mental health clinics in and around Philadelphia.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of major depressive disorder
* Able to read at the 4th grade level or higher
* Willingness to be randomized and participate in research

Exclusion Criteria:

* Current or past diagnosis of schizophrenia, seizure disorder, bipolar disorder, psychotic features, or clinically significant organic pathology
* Significant suicidal risk/ideation requiring immediate referral for more intensive treatment, or specific gesture in the last 6 months
* Current substance abuse or dependence requiring immediate referral to substance abuse program
* Acute medical problem requiring immediate inpatient treatment
* Need for referral to a partial hospitalization program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12-09 (Actual); Study Completion 2014-12-09 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HAM-D) | 6 months

SECONDARY OUTCOMES:
BASIS-24 | 6 months
Beck Depression Inventory - II (BDI-II) | 6 months
Medical Outcomes Study 36-Item Short Form (SF-36) | 6 months
  Measure of general functionality
Quality of Life Inventory (QOLI) | 6 months
Ways of Responding (WOR) | 2 months
Dysfunctional Attitudes Scale (DAS) | 2 months
Psychological Distance Scaling Task (PDST) | 2 months
Self-Understanding of Interpersonal Patterns Scale-Revised (SUIP-R) | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Gibbons, Ph.D., Principal Investigator — University of Pennsylvania; Paul Crits-Christoph, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Connolly Gibbons MB, Gallop R, Thompson D, Luther D, Crits-Christoph K, Jacobs J, Yin S, Crits-Christoph P. Comparative Effectiveness of Cognitive Therapy and Dynamic Psychotherapy for Major Depressive Disorder in a Community Mental Health Setting: A Randomized Clinical Noninferiority Trial. JAMA Psychiatry. 2016 Sep 1;73(9):904-11. doi: 10.1001/jamapsychiatry.2016.1720. PMID 27487573
- [Derived] Connolly Gibbons MB, Mack R, Lee J, Gallop R, Thompson D, Burock D, Crits-Christoph P. Comparative effectiveness of cognitive and dynamic therapies for major depressive disorder in a community mental health setting: study protocol for a randomized non-inferiority trial. BMC Psychol. 2014 Nov 11;2(1):47. doi: 10.1186/s40359-014-0047-y. eCollection 2014. PMID 25566391